CLINICAL TRIAL: NCT00972296
Title: Comparison of Two Types of Ankle Braces in the Management of Ankle Pain in Hemophilia
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, David Oleson, Principal Investigator, Oregon Health and Science University
Other Study IDs: DOleson
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Arthropathy Due to Bleeding From Hemophilia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Persons with hemophilia with ankle pain
  Interventions: Device: Carbon fiber ankle foot orthosis versus cast boot

INTERVENTIONS:
Device: Carbon fiber ankle foot orthosis versus cast boot — Relief of ankle pain and normalizing of gait using either device.

SUMMARY:
This project proposes to examine the difference in effectiveness of fracture boots and carbon fiber braces in the management of gait abnormalities and pain relief due to ankle pain from arthritis due to ankle bleeds. Fracture boots are "walking casts" that you can put on and take off. They prevent the ankle from moving and have a curved sole to mimic normal walking. They can help relieve pain of ankle arthritis from ankle bleeds by stopping ankle motion and absorbing some of the body's own weight while walking. Carbon fiber braces use newer technology resulting in lighter and smaller braces. They are designed to assist with helping clear the toe and straighten the knee while walking.

Gait analysis wearing both the fracture boot and carbon fiber brace will be performed by walking on a mat equipped with pressure sensors and will examine the effect of the fracture boot and the carbon fiber brace on how you walk. These tests will be compared to walking on the mat without either brace. The sensors on the mat will measure different aspects of gait such as step length and foot position. You will be asked questions about how much ankle pain you have using no brace compared to each brace.

People with hemophilia A or B and ankle pain from bleeds will be asked to participate. They will be approached during routine clinic visits and will also be contacted by telephone.

Levels of pain will be measured before, during and after each trial using standardized visual analog and ordinal pain scales. Measurements from the gait mat and levels of pain relief will be used to determine effectiveness of each type of support.

Statisticians will be used to analyze results of the gait mat and pain scale measurements.

ELIGIBILITY:
Inclusion Criteria:

* Hemophilia A or B, with or without inhibitor, with unilateral or bilateral ankle pain

Exclusion Criteria:

* None

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients followed at the Oregon Hemophilia Treatment Center
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Pain relief measured by lower pain score with either AFO or cast boot | Outcome to be assessed at the time of trial

SECONDARY OUTCOMES:
Improvement of gait parameters | To be assessed at time of trial

CONTACTS AND LOCATIONS:
Locations (1):
- Child Development and Rehabilitation Center, Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] 1. Bladen M, Alderson L, Khair K, Liesner R, Green J, Main E. Can early subclinical gait changes in children with haemophilia be identified using the GAITRite® walkway, Haemophilia; Sep2007, Vol. 13 Issue 5, p542-547 2. Wall J, Bruni B, Chapter 17, Clinical Gait Analysis: Temporal and Distance Parameters, Assessment in Occupational Therapy and Physical Therapy, edited by J.V. Van Deusen, 1996